CLINICAL TRIAL: NCT01993667
Title: Acetazolamide for the Prevention of High Altitude Illness: a Comparison of Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Scott McIntosh, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50402
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Prophylaxis of Acute Mountain Sickness
MeSH Terms: interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetazolamide normal dose (Active Comparator): Experimental : Acetazolamide 125 mg twice daily
  Interventions: Drug: Normal Dose Acetazolamide
- Acetazolamide low dose (Experimental): Experimental: Acetazolamide 62.5 mg twice daily
  Interventions: Drug: Low Dose Acetazolamide

INTERVENTIONS:
Drug: Low Dose Acetazolamide — Administration of low dose acetazolamide
  Other Names: Diamox
  Arms: Acetazolamide low dose
Drug: Normal Dose Acetazolamide — Administration of normal dose acetazolamide
  Other Names: Diamox
  Arms: Acetazolamide normal dose

SUMMARY:
This is a phase 4, randomized, double-blinded interventional trial comparing alternative doses of Acetazolamide for the prevention of High Altitude Illness.

DETAILED DESCRIPTION:
Acetazolamide, or Diamox, is the standard medical prophylaxis agent for high altitude illness. The medication is effective in preventing acute mountain sickness (AMS), high altitude pulmonary edema (HAPE), and high altitude cerebral edema (HACE). Its mechanism is via inhibition of the carbonic anhydrase enzyme which counteracts the respiratory alkalosis which occurs during ascent to altitude. It facilitates the excretion of bicarbonate in the urine. As a result, acetazolamide hastens acclimatization and helps prevent high altitude disorders.

Current recommended dosing is 125 mg, orally twice daily, started 24 hours prior to ascending in elevation. Side effects include tingling of the fingers and toes and perioral numbness which may be erroneously interpreted as stroke symptoms. Since acetazolamide is a mild diuretic, frequent micturition may occur leading to interruption of daytime activities as well as broken sleep. These effects can affect safety at high altitude. Acetazolamide is normally discontinued 2 days after the user has reached their highest elevation or a plateau in elevation.

A lower dose may be just as effective in preventing high altitude illnesses while preventing the disconcerting side effects resulting from its use. A smaller dose has not been studied, however. We will compare the common dose of 125 mg twice daily with a lower dose of 62.5 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English or Indian speaking
* Mountaineers or trekkers who plan to climb Mt. McKinley or trek to Base Camp on Mt. Everest

Exclusion Criteria:

* Low sodium and/potassium blood serum levels
* Kidney disease or dysfunction
* Liver disease, dysfunction, or cirrhosis
* Suprarenal gland failure or dysfunction
* Hyperchloremic acidosis
* Angle-closure glaucoma
* Taking high dose aspirin (over 325 mg/day)
* Any reaction to sulfa drugs or acetazolamide
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McIntosh Scott, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetazolamide Normal Dose: Experimental : Acetazolamide 125 mg twice daily
  Acetazolamide: Administration of low dose acetazolamide
- Acetazolamide Low Dose: Experimental: Acetazolamide 62.5 mg twice daily
  Acetazolamide: Administration of low dose acetazolamide
Period: Overall Study
Arm/Group | Acetazolamide Normal Dose | Acetazolamide Low Dose
Started | 64 | 66
Completed | 43 | 47
Not Completed | 21 | 19
Not completed — Insufficient data to analyze | 16 | 16
Not completed — Insufficient altitude reached | 3 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide Normal Dose | Acetazolamide Low Dose | Total
Number analyzed (Participants) | 43 | 47 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (12.7) | 41.6 (13.5) | 43.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Mountain Sickness as Measured by the Lake Louise Score
Description: Lake Louise Score, A total score of 3 to 5 indicates mild AMS. A score of 6 or more signifies severe AMS. Minimum value - 0, Maximum = 15
Time Frame: 12 days
Population: Seventy-three participants had sufficient data to be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide Normal Dose | Acetazolamide Low Dose
Number analyzed (Participants) | 35 | 38
Participants | 21 | 21

2. Secondary Outcome: Number of Participants With Side Effects
Description: The typical side effects of acetazolamide will be measured daily (paresthesias of fingers and toes, change in urination frequency, and change in taste of beverages).
  The side effect questionnaire included the following questions: In the past 12 h, have you experienced the following symptoms: Tingling of toes? Tingling of fingers? Increase in urination? Taste change of beverages? Symptoms were self-reported and rated on a 0-5 scale (0=none, 5=maximum)
Time Frame: 12 days
Population: These participants had sufficient data to be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetazolamide Normal Dose | Acetazolamide Low Dose
Number analyzed (Participants) | 35 | 38
Participants | 6 | 7

ADVERSE EVENTS:
Time Frame: 12 days
Arm/Group | Acetazolamide Normal Dose | Acetazolamide Low Dose
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/47
Other Adverse Events (participants affected / at risk) | 0/43 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No